CLINICAL TRIAL: NCT01930448
Title: Mechanisms of Diabetes Control After Weight Loss Surgery, Sub-study #1
Status: Withdrawn | Type: Observational
Why Stopped: PI relocated to another Institution
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 03-108
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Gastric Bypass Surgery; Gastric Banding; Type 2 Diabetes
Keywords: Bariatric; Gastric Bypass; Gastric Banding,; Type 2 Diabetes; Incretins; GLP-1; GIP; Insulin secretion; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- gastric bypass: Surgical group of obese patients with type 2 diabetes undergoing gastric bypass surgery
- gastric banding: surgical group of obese patients with type 2 diabetes undergoing gastric banding

SUMMARY:
Gastric bypass (GBP) and laparoscopic adjustable banding (AGB) are common procedures that can result in significant weight loss and significantly improve type 2 diabetes in 40-80% of cases. The mechanism and time course of these changes have not been well studied and are poorly understood. The primary aim of this study is to investigate the potential weight-independent mechanisms of diabetes remission after GBP, by comparing GBP and AGB subjects after similar weight loss.

DETAILED DESCRIPTION:
All participants will be tested before and then after 10 and 20-30% weight loss after either GBP or AGB surgery. Subjects will undergo an oral glucose tolerance test (OGTT) an isoglycemic intravenous glucose test (IVGT) to assess the incretin effect, a measure of insulin sensitivity by an intravenous insulin sensitivity test (IVGTT) and body composition measurements.

ELIGIBILITY:
Inclusion Criteria:

* obese type 2 diabetes individuals scheduled to undergo bariatric surgery by either gastric banding or gastric bypass surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: severly obese patients with type 2 diabetes undergoing gastric bypass or gastric banding
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Incretin Effect | Before surgery, 1, 12, and 24 months post
  Effect of GBP and AGB on incretin hormones glucagon-like peptide-1 (GLP-1) and gastric inhibitory peptide (GIP)

SECONDARY OUTCOMES:
Change in Body Composition | Before surgery, 12, and 24 months post
  Body composition measurements to determine body volume, size, and fat

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — New York Obesity Nutrition Research Center
Locations (1):
- St. Luke's Roosevelt Hospital-New York Obesity Nutrition Research Center, New York, New York, United States